CLINICAL TRIAL: NCT01778543
Title: Pathogenesis and Genetics of Microphthalmia, Anophthalmia and Uveal Coloboma ( MAC)
Brief Title: Pathogenesis and Genetics of Microphthalmia, Anophthalmia and Uveal Coloboma (MAC)
Status: Recruiting | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130049; 13-EI-0049
Record Dates: First submitted 2013-01-26; First posted 2013-01-29 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-09-30

CONDITIONS: Coloboma; Anophthalmia; Microphthalmia
Keywords: Repository; Natural History; Genetics
MeSH Terms: conditions — Coloboma; Anophthalmos; Microphthalmos

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MAC: Participants with MAC and their family members.

SUMMARY:
Background:

- Uveal coloboma is a condition where the eye does not form normally. It occurs early in the fetus s development during pregnancy. It can lead to different kinds of eye problems, including blindness. Uveal coloboma is part of a spectrum of developmental eye conditions that include anophthalmia and microphthalmia, typically referred to as "MAC". Several genes have been linked to MAC, but the cause of most causes are hard to find. Researchers want to study the genes of people who have MAC and genes from their close, unaffected relatives (such as parents and siblings).

Objectives:

- To study the genes associated with MAC.

Eligibility:

- Individuals at least 1 years of age who either have MAC or are an unaffected relative (such as a parent or sibling).

Design:

* Participants will have a physical exam and medical history. They will also have a full eye exam.
* Participants with MAC may have other exams, such as imaging studies and hearing assessments.
* All participants will also provide blood, cheek swab or saliva or DNA samples for genetic testing.

DETAILED DESCRIPTION:
Objective: The objectives of this study are to: 1) define ocular, systemic, and other associations in a cohort of well-phenotyped participants with microphthalmia, anophthalmia and/or uveal coloboma (MAC); 2) define risk factors and microforms of MAC in relatives of affected individuals; and 3) establish a repository of DNA and/or lymphoblastoid cell lines from select participants for use in laboratory investigations when scientifically indicated.

Study Population: Six hundred (600) individuals of at least one year of age with documented MAC and their relatives will be enrolled. A subset of approximately 100 participants who are eligible and interested will be referred to enroll in this study from the Microphthalmia, Anophthalmia, and Coloboma Genetic Epidemiology in Children (MAGIC Study) at Baylor College of Medicine (Baylor Protocol # H-49046, NCT06293560).

Design: This is a natural history/genetic repository study. Six hundred (600) participants will be enrolled over fifteen years. Participants will undergo a complete age-appropriate baseline eye examination and physical examination and provide a blood, buccal cell/saliva, or DNA sample.

Outcome Measures: The tests, data and samples collected will be analyzed to better understand the genetics of MAC. In particular, ocular, and systemic associations will be defined in a cohort of well-phenotyped participants with MAC, as will the risk factors and microforms of these disorders in relatives of affected individuals.

ELIGIBILITY:
* INCLUSION CRITERIA:
* The participant must be one year of age or older.
* The participant must be able to cooperate with an age-appropriate eye examination or be able to provide a copy of a complete eye examination report.
* The participant must be able to provide a blood, buccal/saliva, or DNA sample.
* The participant must be able to understand and sign this protocol s informed consent form OR have a legal parent/guardian/representative with the ability to do the same.
* The participant must either:

  * a. be affected by MAC(i) OR
  * b. be an asymptomatic relative of an affected individual.

    (i) Participants will be considered to be affected if they have a clear ocular phenotype related to MAC or if they are deemed affected by other clinical evaluations (e.g., the presence of a unique, systemic manifestation co-segregating with MAC, or a rare or unique kidney finding).

EXCLUSION CRITERIA:

* Female participants who are pregnant are not eligible for enrollment. After giving birth, the female participant and/or a legal parent/guardian/representative may reach out regarding participation in the study.
* Participants who are NEI employees or subordinates or co-workers of an investigator will be excluded from this study; however, non-NEI NIH employees may enroll in the study.

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be ascertained through other pre-existing protocols, such as the NEI Ocular Natural History protocol (16-EI-0134), the NEI Screening protocol (08-EI-0102), through another similar, existing protocol or through referral from an outside clinician after a review of pertinent medical records. Six hundred (600) participants of at least one year of age with documented MAC and their relatives will be enrolled. A subset of approximately 100 participants who are eligible and interested will be referred to enroll in this study from the MAGIC Study at Baylor College of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2013-01-08 (Actual); Primary Completion 2027-12-27 (Estimated)

PRIMARY OUTCOMES:
The tests, data, and samples collected will be analyzed to better understand the genetics of MAC. | end of study
  The tests, data, and samples collected will be analyzed to better understand the genetics of MAC.

CONTACTS AND LOCATIONS:
Overall Officials: Brian P Brooks, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2013-EI-0049.html